CLINICAL TRIAL: NCT00351273
Title: Phase 3 Trial to Assess the Efficacy of Long-term (6 Months) Combination Antibiotics as a Treatment for Chlamydia-induced Reactive Arthritis
Brief Title: Combination Antibiotic Treatment for Reactive Arthritis Caused by Chlamydia Bacteria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AR053646 (NIH); R21AR053646 (NIH); 1R21AR053646-01 (NIH)
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2016-06

CONDITIONS: Arthritis, Reactive; Reiter Disease
Keywords: Chlamydia
MeSH Terms: conditions — Arthritis, Reactive; Chlamydia Infections | interventions — Doxycycline; Rifampin; Azithromycin; Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azithromycin and Rifampin (Active Comparator): Participants received Azithromycin and Rifampin
  Interventions: Drug: Azithromycin and Rifampin
- Doxycycline and Rifampin (Active Comparator): Participants received Doxycycline and Rifampin
  Interventions: Drug: Doxycycline and Rifampin
- received placebo (Placebo Comparator): Participants received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline and Rifampin — doxycycline 100mg daily; rifampin 300mg daily (both for 6 months)
  Other Names: Atridox and Rifadin
  Arms: Doxycycline and Rifampin
Drug: Azithromycin and Rifampin — Azithromycin 500mg daily for 5 days and then twice weekly; Rifampin 300mg daily (both for 6 months)
  Other Names: Zithromax and Rifadin
  Arms: Azithromycin and Rifampin
Drug: Placebo — Methylcellulose
  Other Names: Placebo effect
  Arms: received placebo

SUMMARY:
Reactive arthritis, also known as Reiter's syndrome, is a form of arthritis that occurs as a reaction to an infection elsewhere in the body. It is characterized by inflammation of the joints, tendons, urogenital tract, and eyes. Pain and swelling in the knees, ankles, and feet are common. This study will determine the effectiveness of antibiotic therapy in treating people with chlamydia-induced reactive arthritis that has lasted for more than 6 months.

DETAILED DESCRIPTION:
The initial infection that causes reactive arthritis is caused by one of two bacteria: Chlamydia trachomatis, which is usually acquired through sexual contact, or Chlamydia pneumoniae, which can cause respiratory infections. Most people recover fully from the initial flare of arthritis symptoms. However, about 20% of people with reactive arthritis experience long-lasting symptoms. In these individuals, the Chlamydia bacteria exist in a persistent metabolically active state within the joint tissue, even years after the initial exposure. The bacteria produce heat shock proteins (HSPs), which are thought to play a key role in the chronic persistent state of Chlamydia and which may stimulate the immune inflammatory response seen in reactive arthritis. This indicates the need for antimicrobial therapy that can reduce Chlamydia's HSP production and block its metabolism. The purpose of this study is to determine the effectiveness of long-term combination antibiotic therapy in treating people with chronic reactive arthritis. The study will use two different combinations of common antibiotics: doxycycline paired with rifampin and azithromycin paired with rifampin.

This study will entail 6 months of treatment followed by 3 months of follow-up. After screening, eligible participants will be randomly assigned to one of three treatment groups: rifampin once a day plus doxycycline twice a day; rifampin once a day plus azithromycin once a day for 5 days, then twice weekly; or placebo. Study visits will occur at baseline and Months 1, 3, 6, and 9. At all visits, participants will undergo an interview, a physical examination, and blood collection. They will also complete a questionnaire related to their symptoms and functional status. At screening and Month 6, a synovial biopsy may be performed. This will involve taking a sample of the tissue that lines the joints.

ELIGIBILITY:
Inclusion Criteria:

* Meet the following European Spondyloarthropathy Study Group Criteria:

  1. inflammatory spinal pain OR
  2. synovitis AND
  3. one or more of the following:

     1. positive family history
     2. urethritis or cervicitis within 1 month prior to onset of arthritis
     3. buttock pain
     4. enthesopathy
     5. sacroiliitis
* Disease duration of at least 6 months
* Negative pregnancy test at study baseline and willing to use an effective method of contraception other than combined oral contraceptives for the duration of the study (for women of childbearing age)

Exclusion Criteria:

* Sensitivity or history of allergic reaction to rifampin, doxycycline, or azithromycin
* Currently taking any medications that may interact with the study medications, specifically rifampin
* Liver transaminases greater than or equal to two times the normal level
* Significant abnormalities in the complete blood count (CBC)
* Pregnant
* Current psoriasis
* Diagnosis of inflammatory bowel disease
* Diagnosis of ankylosing spondylitis
* Previous prolonged exposure to antibiotics (more than 2 weeks) as a potential treatment for reactive arthritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Carter, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Louisiana State University, New Orleans, Louisiana
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carter JD, Valeriano J, Vasey FB. Doxycycline versus doxycycline and rifampin in undifferentiated spondyloarthropathy, with special reference to chlamydia-induced arthritis. A prospective, randomized 9-month comparison. J Rheumatol. 2004 Oct;31(10):1973-80. PMID 15468362
- [Derived] Carter JD, Espinoza LR, Inman RD, Sneed KB, Ricca LR, Vasey FB, Valeriano J, Stanich JA, Oszust C, Gerard HC, Hudson AP. Combination antibiotics as a treatment for chronic Chlamydia-induced reactive arthritis: a double-blind, placebo-controlled, prospective trial. Arthritis Rheum. 2010 May;62(5):1298-307. doi: 10.1002/art.27394. PMID 20155838

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin & Rifampin: Participants will receive Azithromycin and Rifampin
- Doxycycline & Rifampin: Participants will receive Doxycycline and Rifampin
- Placebo: Participants will receive placebo
Period: Overall Study
Arm/Group | Azithromycin & Rifampin | Doxycycline & Rifampin | Placebo
Started | 15 | 12 | 15
Completed | 14 | 10 | 10
Not Completed | 1 | 2 | 5
Not completed — Lost to Follow-up | 1 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin & Rifampin | Doxycycline & Rifampin | Placebo | Total
Number analyzed (Participants) | 15 | 12 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 13 | 40
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12) | 43.8 (12.3) | 49 (16.3) | 45.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 6 | 18
  Male | 8 | 7 | 9 | 24
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 14 | 41
  Canada | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigate Whether a 6 Month Course of Combined Antibiotics Was Effective Treatment.
Description: The outcome measure was a composite endpoint. Participants had to meet 4/6 clinical criteria. 17/24 subjects randomized to combination antibiotics did respond to treatment when compared to 3/10 randomized to placebo.
Time Frame: Month 6
Population: Efficacy and safety analyses were performed on an intent to treat(ITT) basis. Subjects who prematurely withdrew or who were lose to follow up for any reason were included in the ITT population and were considered nonresponders.
Measure: Number; unit: participants
Arm/Group | Azithromycin & Rifampin | Doxycycline & Rifampin | Placebo
Number analyzed (Participants) | 14 | 10 | 10
participants | 10 | 7 | 3
Statistical Analysis 1: Comparison: Azithromycin & Rifampin vs Doxycycline & Rifampin vs Placebo; Difference in the percentages of participants with response between all those who received combination therapy vs. placebo; Test type: Superiority or Other; p = 0.01, Fisher Exact; Mean Difference (Final Values) = 40.8

2. Secondary Outcome: Number of Patients With a Complete Response (Resolution of All Symptoms)
Description: Patients who completed full 6 months of treatment that reported feeling complete resolution of symptoms at month 6 visit and had no worsening of condition at the month 9 follow up visit.
Time Frame: Months 6 and 9
Population: Patients randomized to combination antibiotics who believed that their disease went into complete remission during the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Rifampin | Doxycycline and Rifampin | Received Placebo
Number analyzed (Participants) | 10 | 7 | 3
Participants | 5 | 1 | 0

3. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: Comparison of mean ESR rates of combination antibiotic group vs placebo group at Baseline, Month 1, 3, 6 and 9
Time Frame: Baseline Month 1, 3, 6 and 9
Measure: Mean (Full Range); unit: millimeters/hour
Groups:
- Combination Antibiotic: Group who recieved either combination of antibiotics
- Placebo: Group who recieved placebo
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
millimeters/hour
  Baseline | 25.1 [1 to 81] | 18.9 [1 to 74]
  Month 1 | 17.8 [2 to 50] | 25.2 [1 to 78]
  Month 3 | 17.7 [1 to 72] | 19.8 [4 to 42]
  Month 6 | 12.7 [1 to 55] | 17.0 [3 to 37]
  Month 9 | 14.0 [1 to 47] | 18.4 [4 to 45]

4. Secondary Outcome: hsCRP
Description: Comparison of high sensitivity C-reactive protein measurement in combination antibiotic group vs placebo group at Baseline, Month 1, 3, and 6
Time Frame: Baseline, Month 1, 3, and 6
Measure: Mean (Full Range); unit: mg/litre
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
mg/litre
  Baseline | 1.07 [0.02 to 10.9] | 0.42 [0.069 to 1.85]
  Month 1 | 0.56 [0.02 to 3.65] | 0.27 [0.106 to 0.651]
  Month 3 | 0.63 [0.02 to 5.88] | 0.55 [0.035 to 2.51]
  Month 6 | 0.41 [0.02 to 2.34] | 0.34 [0.02 to 0.796]

5. Secondary Outcome: HAQ DI Score
Description: Comparison of HAQ-DI score of combination antibiotic group vs placebo group at Baseline, Month 1,3,6 and 9 The Health assessment questionnaire disability index (HAQ-DI) is a questionnaire for the assessment of Rheumatoid Arthritis. The questionnaire is a patient reported outcome (PRO) which is usually self-administered by the patient There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2. In addition, if an aide or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made.
  The 8 scores of the 8 sections are summed and divided
Time Frame: Baseline, Month 1,3,6 and 9
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
score on a scale
  Baseline | 0.84 [0 to 3] | 1.1 [0 to 3]
  Month 1 | 0.79 [0 to 3] | 0.92 [0 to 3]
  Month 3 | 0.68 [0 to 3] | 0.87 [0 to 3]
  Month 6 | 0.71 [0 to 3] | 0.99 [0 to 3]
  Month 9 | 0.57 [0 to 3] | 0.92 [0 to 3]

6. Secondary Outcome: PhGA Assessment
Description: Comparison of Physician's global assessment of disease activity (PhGA) using 0-100mm visual analog scale (VAS) , where 0 indicates the best possible outcome and 100 indicates the worst possible outcome, in combination antibiotic vs placebo groups at Baseline, month 1,3,6 and 9
Time Frame: Baseline, month 1,3,6 and 9
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
units on a scale
  Baseline | 63.9 [44 to 91] | 60.2 [3 to 85]
  Month 1 | 35.2 [2 to 70] | 52.9 [24 to 77]
  Month 3 | 23.2 [0 to 51] | 49.4 [5 to 74]
  Month 6 | 16.3 [0 to 49] | 45.7 [0 to 72]
  Month 9 | 17.7 [0 to 50] | 43.8 [2 to 72]

7. Secondary Outcome: Swollen 76 Joint Count (SJC)
Description: Comparison of modified Swollen Joint Counts between combination antibiotic and placebo groups at Baseline, Month 1, 3, 6 and 9. Determination of swelling in each of the 76 joints was determined by any swelling or absence of swelling. Each swollen joint receives a value of 1, ranging from 0-76 as a possible score.
Time Frame: Baseline, month 1,3,6 and 9
Measure: Mean (Full Range); unit: Swollen Joints
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
Swollen Joints
  Baseline | 4.1 [0 to 12] | 4.5 [0 to 9]
  Month 1 | 1.7 [0 to 6] | 3.5 [0 to 8]
  Month 3 | 0.9 [0 to 4] | 4.3 [0 to 13]
  Month 6 | 0.9 [0 to 5] | 5.2 [0 to 13]
  Month 9 | 0.5 [0 to 4] | 5.1 [0 to 12]

8. Secondary Outcome: 78 Tender Joint Count (TJC)
Description: Comparison of modified 78 Tender Joint Count (TJC) between combination antibiotic and placebo groups at Baseline, Month 1, 3, 6 and 9. Determination of tender joing in each of the 78 joints was determined by examination. Each tender joint receives a value of 1, ranging from 0-78 as a possible score.
Time Frame: Baseline, Month 1, 3, 6 and 9
Measure: Mean (Full Range); unit: Tender Joints
Arm/Group | Combination Antibiotic | Placebo
Number analyzed (Participants) | 27 | 15
Tender Joints
  Baseline | 7.4 [1 to 20] | 9.6 [0 to 24]
  Month 1 | 5.0 [0 to 23] | 10.6 [0 to 25]
  Month 3 | 3.3 [0 to 17] | 10.8 [0 to 28]
  Month 6 | 2.0 [0 to 9] | 11.8 [0 to 37]
  Month 9 | 1.9 [0 to 9] | 10.9 [0 to 29]

ADVERSE EVENTS:
Arm/Group | Azithromycin & Rifampin | Doxycycline & Rifampin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No